CLINICAL TRIAL: NCT04234334
Title: Evaluation of the Role of Eggs on Antioxidant Status, Plasma Choline and Lipoprotein Metabolism in Adults With Metabolic Syndrome Consuming a Plant-based Diet
Brief Title: Benefits of Eggs in Combination With a Plant-based Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Maria Luz Fernandez, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H19-178
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease; Diabetes; Metabolic Syndrome
Keywords: eggs; lutein; zeaxanthin; choline; metabolic syndrome; plant-based diet
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Crossover design
Who Masked: Participant
Masking Description: Egg or Egg substitutes (whites only) will be provided to subjects and since they are similar in appearance and color, they will not know when they are consuming them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg intake (Experimental): Consumption of 2 eggs with spinach daily for breakfast for 4 weeks
  Interventions: Other: Consume 2 eggs with spinach per day
- Egg Subsitute (Experimental): Consumption of 2 egg substitutes daily for breakfast for 4 weeks
  Interventions: Other: Egg Subsitute with spinach per day

INTERVENTIONS:
Other: Consume 2 eggs with spinach per day — Participants will be randomly allocated to consume either 2 eggs or 2 egg substitutes with spinach daily for 4 weeks and after a 3-week wash out, they will be allocated to the alternate treatment
  Other Names: Egg substitute
  Arms: Egg intake
Other: Egg Subsitute with spinach per day — Egg Subsitute with spinach per day
  Arms: Egg Subsitute

SUMMARY:
The main objective of the study is to demonstrate that the inclusion of eggs to a plant-based diet will not increase the risk for heart disease but will increase the concentration of lutein and zeaxanthin, two important antioxidants and will also increase choline, an important component of membrane phospholipids.

DETAILED DESCRIPTION:
Results from studies involving cells, animal models and clinical trials have demonstrated that lutein and zeaxanthin potentially protect against chronic diseases, including age-related macular degeneration, cataracts, coronary heart disease and stroke. Plasma concentrations of lutein and zeaxanthin are closely associated with their antioxidant properties and with their protection against reactive oxygen species (ROS).

Choline is recognized as an essential nutrient for health because of its many functions in growth and development, as well as neurological function and formation of membrane phospholipids, including phosphatidylcholine (PC) and sphingomyelin.

Therefore the objective of this study is to demonstrate that inclusion of eggs in a plant-based diet will potentiate the benefits of this healthy diet by increasing plasma concentrations of lutein, zexanthin and choline presents in egg yolks and theoretically increase the antioxidant and anti-inflammatory actions of these components. This would be potentially more important in those individuals with metabolic syndrome, which is the target population of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* 35-70 years
* Metabolic syndrome (based on 3 out of 5 characteristics: waist circumference. 88 cm for women and > 102 cm for men; plasma triglycerides > 150 mg/dL, blood pressure > 135/85 mm Hg, fasting glucose > 100 mg/dL and HDL < 40 mg/dL for men and < 50 mg/dL for women)
* Willing to consume a spinach omelet made with 2 eggs or the equivalent amount of egg substitute daily for 4 weeks each
* Willing to follow a plant-based diet for 13 weeks
* Not have cardiovascular disease, high cholesterol, diabetes, cancer, liver or renal disease
* Proficient in English

Exclusion Criteria:

* Self-reported diabetes, cardiovascular disease, history of stroke, liver disease or cancer
* Taking glucose lowering medications
* Triglycerides > 500 mg/dL
* Cholesterol > 240 mg/dL
* Blood pressure > 145/100 mm Hg
* Allergic to eggs or spinach

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Plasma lutein | 1 year
  Plasma lutien will be measured by HPLC. The units are expresses as µmol/L
Plasma choline | 1 year
  It will be measured by mass spectometry. The units are expressed as nmol/mL
Plasma Zeaxanthin | 1 year
  Plasma zeaxanthin will by measured by HPLC. The units are expressed as µmol/L

SECONDARY OUTCOMES:
Plasma lipids | 1 year
  Total, LDL and HDL cholesterol and triglycerides will be measured by an automated spectrometer simultaneously. The units are expressed as mg/dL
Plasma glucose | 1 Year
  Plasma glucose will be measured by an automated spectrometer. Units are expressed as mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Luz Fernandez, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Department of Nutritional Sciences, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No